CLINICAL TRIAL: NCT05162508
Title: Characterization of the Impact of SARS-CoV-2 Variability on the Course of COVID-19 in Patients With Severe Disease Hospitalized in Intensive Care Units: Prospective Observational Multicentric Study
Brief Title: Impact of COVID-19 SARS-CoV-2 Variability in ICU Hospitalized Patients With Severe Disease
Acronym: SEVARVIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211494
Record Dates: First submitted 2021-12-10; First posted 2021-12-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-08

CONDITIONS: SARS-CoV2 Infection; COVID-19 Acute Respiratory Distress Syndrome; Mutation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nasopharyngeal swab — Nasopharyngeal swab available in Standard Of Care (SOC) will be analysed (Full-length SARS-CoV-2 RNA sequencing and Transcriptomic analyses)

SUMMARY:
Background:The impact of the emergence of SARS-CoV-2 variants on the severity and clinical outcomes of COVID-19 is controversial. Whether virological characteristics including the mutational patterns of the different viral proteins (e.g., Spike, NSP proteins, ORF6) could be associated with a different immune response and subsequent severity of the disease is unknown. ln the next coming months, new variants carrying the same or new mutational patterns will continue to emerge. Monitoring their dynamics over time and their impact on disease severity is required for refining national and international disease control policies.

Main objective: To unravel the relationships between specific viral mutations/mutational patterns and the clinical outcomes of COVID-19 in patients hospitalized in intensive care units (ICUs) for acute respiratory failure following severe SARS-CoV-2 infection.

Design of the study Prospective multicentre observational cohort study

Schedule for the study: Inclusion period: 24 months; Participation period: 28 days ; Total duration : 24 months + 28 days;

DETAILED DESCRIPTION:
Background:The impact of the emergence of SARS-CoV-2 variants on the severity and clinical outcomes of COVID-19 is controversial. Preliminary studies estimated that the probability of death associated with variant of concern (VOC) B.1.1.7, the UK variant, is 55% higher than that associated with pre-existing variants. However, no difference has been found in another study. In Brazil, infection with VOC P1 has been suggested to be associated with an increased case fatality rate in young adults. The effect of other "variants of concern" (Beta, B.1.351; Delta, B.1.617.2, or the most recent Omicron variants) or "variants of interest" (A27, B.1.525, etc.) on the severity of the disease and the prognosis of severe forms is unknown. More generally, whether virological characteristics including the mutational patterns of the different viral proteins (e.g., Spike, NSP proteins, ORF6) could be associated with a different immune response and subsequent severity of the disease is unknown. ln the next coming months, new variants carrying the same or new mutational patterns will continue to emerge in different geographic areas, as a result of the collective immune pressure induced by natural infection and vaccination. Monitoring their dynamics over time and their impact on disease severity is required for refining national and international disease control policies.

In this project, a large prospective multicenter observational cohort promoted by the Assistance Publique-Hôpitaux de Paris (AP-HP) will be conducted, to understand the effect of SARS-CoV-2 genetic variability on the outcome of COVID-19 disease in patients with severe illness. The study will include critically ill patients hospitalized for acute respiratory failure/acute respiratory distress syndrome (ARDS) associated with COVID-19. The objective of the work will be to characterize the SARS-CoV-2 variants found in this population over time, and to identify and phenotypically characterize specific mutations/mutational patterns associated with the different clinical outcomes (primary clinical endpoint defined as mortality at day-28). The impact of the mutations on viral infectivity, sensitivity to neutralizing antibodies and ability to induced cytokine production will be assessed in vitro and ex-vivo respectively, in appropriate models available in the laboratory. Further to full-length viral genome sequencing, our in-house shotgun metagenomics method will be used to characterize the effect of SARS-CoV-2 variations on respiratory transcriptomic expression profiles and the relationship with the clinical evolutionary profiles.

Design of the study Prospective multicentre observational cohort study

Main objective: To unravel the relationships between specific viral mutations/mutational patterns and the clinical outcomes of COVID-19 in patients hospitalized in intensive care units (ICUs) for acute respiratory failure following severe SARS-CoV-2 infection.

Schedule for the study: Inclusion period: 24 months; Participation period: 28 days ; Total duration : 24 months + 28 days;

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Availability of nasopharyngeal swab from SOC
* SARS-CoV-2 infection as assessed by a positive RT-PCR test (CT < 32), including in SARS CoV-2 vaccinated or previously infected patients
* Patient admitted in the ICU for acute respiratory failure (SpO2 ≤ 90% and need for supplemental oxygen or any kind of ventilator support; i.e., OMS 10-category ordinal scale ≥5)
* Patient or trusted person or close or relative, And, accepting study participation

Exclusion Criteria:

* Patient with SARS-CoV-2 infection but no acute respiratory failure
* Patient deprived of liberty or under legal protection (guardianship, curators, legal protection, forced hospitalization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe SARS-CoV-2 infection and acute respiratory failure admitted in one of the participating ICUs during 2 years of inclusion period.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Day-28 vital status | at Day-28 after admission in intensive care units (ICUs) for acute respiratory failure following severe SARS-CoV-2 infection
  vital status (living / deceased)

CONTACTS AND LOCATIONS:
Overall Officials: Slim FOURATI, MD-PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP) Henri Mondor
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No
AP-HP is the owner of the data. The data cannot be used or disclosed to a third party without its prior permission

REFERENCES:
- [Derived] Audureau E, Bay P, Preau S, Favory R, Guigon A, Heming N, Gault E, Pham T, Chaghouri A, Turpin M, Morand-Joubert L, Jochmans S, Pitsch A, Meireles S, Contou D, Henry A, Roux D, Le Hingrat Q, Kimmoun A, Hartard C, Pene F, L'Honneur AS, Guillon A, Handala L, Tamion F, Moisan A, Daix T, Hantz S, Delamaire F, Thibault V, Darreau C, Thomin J, Pawlotsky JM, Fourati S, de Prost N; SEVARVIR investigators. Clinical Phenotypes of Critically Ill Patients with COVID-19 Infected with Omicron: A Nationwide Prospective Cohort Study. Infect Dis Ther. 2026 Feb;15(2):605-628. doi: 10.1007/s40121-025-01291-3. Epub 2026 Jan 6. PMID 41493514